CLINICAL TRIAL: NCT03354377
Title: A Nutrition-Based Approach to Reduce Heart Disease Risk Among Overweight African Americans: Use of Soul Food Plant-Based or Omnivorous Diets to Address Cardiovascular Disease
Brief Title: Nutritious Eating With Soul (The NEW Soul Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00064855
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Cardiovascular Disease Risk Factors; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan Diet (Experimental): Participants in this group will follow a plant-based vegan diet. The vegan group diet will be based on investigators' pilot work, which instructs participants to favor a diet built around whole grains, fruits, vegetables, and legumes. This group will be supplemented by the Oldways African Heritage and Health program, which includes a food pyramid guide. A Taste of African Heritage (ATAH) six-lesson nutrition and cooking program and an online course for health professionals and cooking instructors (all research and restaurant team members will complete this course.
  Interventions include intervention meetings, physical activity, and podcasts/mailings.
  Interventions: Behavioral: Dietary Intervention Meetings; Behavioral: Physical Activity; Behavioral: Podcasts/Mailings
- Omnivorous (Omni) Diet (Experimental): Participants in this group will follow a low-fat omni diet. The diet intervention for the omni group will be supplemented by the Oldways African Heritage and Health program, which includes a food pyramid guide, A Taste of African Heritage (ATAH) six-lesson nutrition and cooking program and an online course for health professionals and cooking instructors (all research and restaurant team members will complete this course).
  Interventions include intervention meetings, physical activity, and podcasts/mailings.
  Interventions: Behavioral: Dietary Intervention Meetings; Behavioral: Physical Activity; Behavioral: Podcasts/Mailings

INTERVENTIONS:
Behavioral: Dietary Intervention Meetings — Participants will attend classes once per week for the first 6 months, bi-weekly for the next 6 months; then once a month for the last 12 months.
Behavioral: Physical Activity — Participants will be given the following exercise recommendations: strength training twice per week and ≥75 min of vigorous or ≥150 min of moderate PA per week and will be provided with accelerometers.
Behavioral: Podcasts/Mailings — Participants with receive additional support delivered remotely months 13-24 in the form of audio podcasts and email newsletters.

SUMMARY:
This study addresses two challenges seen among African American (AA) participants during previous weight loss and dietary interventions aimed at reducing cardiovascular disease (CVD) risk: poor weight loss results and high attrition rates. Investigators will target both of these challenges by using a randomized design to compare a plant-based dietary intervention (vegan diet) vs. an omnivorous (omni) diet and by focusing on culturally-tailored food choices for AA adults living in the South. Therefore, the objective of the study is to conduct a culturally-tailored, randomized trial examining how a vegan diet affects CVD risk factors and weight as compared with an omni diet. The study will randomize overweight AA adults (n=130) to follow one of two different diets (vegan or omni) for 24 months. Investigators will accomplish objectives and test hypotheses by following two specific primary aims:

Primary Aims: Using a randomized design, determine the impact at 12 months of two different, culturally tailored diets (n=65 omni and n=65 vegan) on changes in:

1. Risk factors for CVD, including LDL cholesterol and blood pressure; and
2. Body weight.

   Secondary Aim
3. Examine long-term changes in CVD risk factors and body weight at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American
* Be between the ages of 18-65 years
* Body Mass Index between 25- 49.9 kg/m2
* Live in the Columbia, SC/Midlands area
* Be able to attend all monitoring and weekly class visits
* Be willing to be randomized to either diet

Exclusion Criteria:

* Currently following a vegan diet
* Diagnosed with diabetes that is controlled by medication
* Currently pregnant or breastfeeding (or plan to become pregnant in the next 24 months)
* Under the age of 18 years old
* Over the age of 65 years old
* Currently participating in a weight loss program
* Has lost more than 10 pounds in the past 6 months
* Diagnosed with stroke or heart attack

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Disease Prevention based on dietary approach. | Two years
  Which dietary approach (vegan or omni) best targets both cardiovascular disease prevention and weight loss among overweight African Americans.

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, PhD, MS, RD, Principal Investigator — University of South Carolina
Locations (1):
- Discovery, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turner-McGrievy GM, Wilcox S, Frongillo EA, Murphy EA, Kim Y, Hu EA, Okpara N, Bailey S. Impact of diet adherence on weight and lipids among African American participants randomized to vegan or omnivorous diets. Obes Sci Pract. 2024 Sep 27;10(5):e70009. doi: 10.1002/osp4.70009. eCollection 2024 Oct. PMID 39345782
- [Derived] Turner-McGrievy GM, Wilcox S, Frongillo EA, Kim Y, Okpara N, Wilson M. Differences in dietary acceptability, restraint, disinhibition, and hunger among African American participants randomized to either a vegan or omnivorous soul food diet. Appetite. 2024 May 1;196:107280. doi: 10.1016/j.appet.2024.107280. Epub 2024 Feb 17. PMID 38373534
- [Derived] Bernhart JA, Quattlebaum M, Eustis S, Okpara N, Wilson MJ, Sentman C, Turner-McGrievy GM. "It's Gonna Be Okay"-A Qualitative Exploration of the COVID-19 Pandemic's Effects on African American Participants During a Dietary Intervention Study. J Acad Nutr Diet. 2023 Dec;123(12):1763-1771. doi: 10.1016/j.jand.2023.07.003. Epub 2023 Jul 16. PMID 37437808
- [Derived] Turner-McGrievy GM, Wilcox S, Frongillo EA, Murphy EA, Hutto B, Wilson M, Davey M, Bernhart JA, Okpara N, Bailey S, Hu E. Effect of a Plant-Based vs Omnivorous Soul Food Diet on Weight and Lipid Levels Among African American Adults: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2250626. doi: 10.1001/jamanetworkopen.2022.50626. PMID 36633848
- [Derived] Bernhart JA, Fellers AW, Wilson MJ, Hutto B, Bailey S, Turner-McGrievy GM. COVID-19 Pandemic Associations on Mental and Physical Health in African Americans Participating in a Behavioral Intervention. J Racial Ethn Health Disparities. 2023 Dec;10(6):3070-3076. doi: 10.1007/s40615-022-01481-6. Epub 2022 Dec 5. PMID 36469289
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 Aug 21;8(8):CD011737. doi: 10.1002/14651858.CD011737.pub3. PMID 32827219
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 May 19;5(5):CD011737. doi: 10.1002/14651858.CD011737.pub2. PMID 32428300